CLINICAL TRIAL: NCT03237611
Title: Phase II Trial Testing the Antiemetic Efficacy of a Single-day Low Dose Aprepitant (or Fosaprepitant) Added to a 5-HT3 Receptor Antagonist Plus Dexamethasone in Patients Receiving Carboplatin
Brief Title: Low Dose Aprepitant for Patients Receiving Carboplatin
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Expired IRB approval on 2/11/21
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Jacobi Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-5109
Record Dates: First submitted 2017-07-31; First posted 2017-08-02 (Actual); Results first posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
Keywords: emesis; aprepitant; carboplatin; chemotherapy-induced nausea and vomiting
MeSH Terms: conditions — Vomiting | interventions — Aprepitant; fosaprepitant; Dexamethasone; Ondansetron

STUDY DESIGN:
Intervention Model Description: Patient scheduled for the first cycle of carboplatin-based chemotherapy will be offered to receive 125mg of oral aprepitant or 115mg of fosaprepitant intravenously for prevention of chemotherapy-induced nausea and vomiting
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- low dose aprepitant or fosaprepitant (Experimental): In addition to standard prophylactic antiemetics (Ondansetron 16mg and Dexamethasone 20mg) patients will be given aprepitant 125mg orally or 115mg fosaprepitant intravenously prior to the first cycle of carboplatin-based chemotherapy. No medications will be given afterwards
  Interventions: Drug: Aprepitant 125 mg; Drug: Fosaprepitant 115 MG; Drug: Dexamethasone; Drug: Ondansetron 16 MG

INTERVENTIONS:
Drug: Aprepitant 125 mg — Patient scheduled for the first cycle of carboplatin-based chemotherapy will be offered to receive low doses of aprepitant (125mg of oral aprepitant) or 115mg of fosaprepitant intravenously for prevention of chemotherapy-induced nausea and vomiting
Drug: Fosaprepitant 115 MG — Patient scheduled for the first cycle of carboplatin-based chemotherapy will be offered to receive low doses of aprepitant (125mg of oral aprepitant) or 115mg of fosaprepitant intravenously for prevention of chemotherapy-induced nausea and vomiting
Drug: Dexamethasone — Dexamethasone will be given as a part of standard CINV prophylaxis for patients receiving carboplatin-based chemotherapy, dosed at 20mg on day 1 of chemotherapy
Drug: Ondansetron 16 MG — Ondansetron will be given as a part of standard CINV prophylaxis for patients receiving carboplatin-based chemotherapy, dosed at 16mg on day 1 of chemotherapy

SUMMARY:
This study evaluates a simple one day prophylaxis of nausea and vomiting for patients who are getting carboplatin based chemotherapy. In addition to standard oral Dexamethasone and oral Ondansetron, participants will be given a third neurokinin 1 (NK1) antagonist agent, either a single dose of oral Aprepitant or intravenous (IV) Fosaprepitant (they have been shown to be equally effective) to improve prevention of nausea and vomiting. No medications need to be taken beyond day 1.

DETAILED DESCRIPTION:
Main predictive factor for the development of Chemotherapy-induced Nausea and Vomiting (CINV) is the emetic potential of a given chemotherapeutic agent. Carboplatin causes both acute and delayed emesis. Guideline groups have typically classified this agent as moderately emetic (MEC); however, its risk of inducing vomiting is at the upper range of this classification, and borders on highly emetic. The recommendation for prevention has been the use of a two-drug regimen (a 5-hydroxytryptamine receptor antagonist (5-HT3RA) plus dexamethasone). The recent randomized studies have shown that patients given only a 2-drug regimen have about a 50% likelihood of emesis if they are women, and about a 30% likelihood of emesis if they are men. Major improvements were reported when a neurokinin-1 receptor antagonist (NK1RA) Aprepitant was added. This improvement is of a similar magnitude to that seen in patients receiving cisplatin. Similar improvements were also seen in a trial in which the NK1RA antiemetic was Rolapitant rather than Aprepitant. The Tanioka and Yahata studies were conducted entirely in patients with gynecologic (GYN) malignancies, and it is not surprising that the control rates are lower in these all female groups.

The most commonly used NK1RA, Aprepitant, is generally given over 3 days. Most studies indicate that this class of agent gives similar results when given in just one day, or over multiple days. Recent studies conducted by Roila compared the efficacy of Aprepitant on day 1 at a low dose (125 mg) versus the full three day regimen totaling 285 mg in patients receiving either cisplatin or the combination of anthracyclines plus cyclophosphamide (AC). In both studies, those patients randomly assigned to just one day of lower dose Aprepitant had control of emesis equal to those receiving multiple days. In both of these trials, patients assigned to the single day Aprepitant arm also received additional antiemetics on days 2 and 3. However, recent studies have failed to show an advantage for continuing dexamethasone after day 1 in patients receiving AC (14) or in those receiving cisplatin. Additionally, a meta-analysis indicated that as long as dexamethasone is given on day 1, there is no advantage to adding a serotonin antagonist (such as ondansetron) after day 1, and ondansetron has been shown to be similar to metoclopramide in the delayed emesis phase. Similarly to studies conducted by Roila, Grunberg and colleagues showed non-inferiority of single-dose intravenous (IV) fosaprepitant (a phosphorylated analog of Aprepitant that is rapidly converted to Aprepitant after IV administration) in a randomized study of patients receiving cisplatin chemotherapy. Fosaprepitant 115 mg IV has been approved as an alternative to the 125-mg oral Aprepitant dose on day 1 of a 3-day regimen.

There is very little data regarding the efficacy of continued steroids after day 1 in patients receiving carboplatin. Recent trials fail to show benefit for continuing dexamethasone after the day of chemotherapy. Aapro and colleagues in a 300 patient trial, showed that dexamethasone in combination with a 5-HT3RA on day 1 gave similar CINV protection to a multiple-day dexamethasone. Similarly, a Japanese study showed no difference in antiemetic efficacy of a single day dexamethasone regimen when prospectively compared with a 3 day dexamethasone regimen; however, the 1 day regimen found significant reductions in steroid induced side effects. Additionally, a large multinational trial in patients receiving AC chemotherapy showed that a single dose of dexamethasone on day 1 along with a single day of NEPA (combination of 5-HT3RA palonosetron with NK1RA Netupitant) offers convenient single-day prophylaxis for both acute and delayed CINV.

Guideline groups are now starting to recommend a 3-agent preventive antiemetic regimen for patients receiving carboplatin, based on the evidence from the studies discussed above. However, not all guideline groups have yet made this recommendation. If it can be shown that a less expensive, more convenient (1-time administration), and potentially safer regimen performs in the same way for patients receiving carboplatin as it did for those receiving cisplatin or AC chemotherapy, and similarly to those receiving 3 days of Aprepitant with carboplatin in the recent randomized trials, a new standard may be established.

Objectives. Primary: To determine in patients receiving their first cycle of carboplatin-based chemotherapy, the complete control rate of emesis (acute and delayed; no vomiting and no use of rescue medications) with the addition of one dose of the oral Aprepitant or intravenous fosaprepitant to a combination of oral dexamethasone + an oral 5-HT3RA (ondansetron).

Secondary: To estimate the control rate on the second cycle of this chemotherapy in those patients agreeing to be assessed in the subsequent chemotherapy cycle.

Methods. CINV will be assessed by using the validated Multinational Association of Supportive Care in Cancer (MASCC) Antiemesis Tool (MAT), which efficiently evaluates the incidence of vomiting and the severity of nausea and vomiting in the acute and delayed emesis periods. Patients will be enrolled at Montefiore Medical Center and at Jacobi Medical Center. Patients will be asked to sign an informed consent form. Patients will be called on day 2 and 5 to remind about form completion, and will return the MAT form on their next outpatient visit (or immediately after completion if the patient is an inpatient). Consent forms then will be kept at a clinical trial center in a file. Case report forms were developed to capture data relevant to research.

Antiemetic Medication administration. Serious adverse events are not expected since a lower dose and frequency of FDA approved medications will be given. They may be obtained or dispensed either by the Jacobi Medical Center, or the Montefiore Medical Center pharmacies, or Aprepitant may be obtained by prescription from an outside pharmacy. If Aprepitant is obtained at an outside pharmacy, the patient will bring the agent to their chemotherapy appointment; all NK1RA drug administration will be directly observed. The use of either Aprepitant or fosaprepitant will be entirely the choice of the ordering oncologist, as both agents are equivalent. Ideally all drugs will be given immediately before (within 5 minutes) chemotherapy; however if a delay occurs up to 2 hours between the antiemetics and chemotherapy, this will be allowable and no additional dosing will be needed. The time of administration of the NK1RA in relation to the chemotherapy will be recorded.

All patients will be given a single dose of 125 mg of Aprepitant orally or 115 mg IV of fosaprepitant prior to the first cycle of carboplatin-based chemotherapy.

Antiemetic drug doses and schedules (same doses in all age and gender groups). Aprepitant or Fosaprepitant: 125 mg of Aprepitant orally immediately prior to chemotherapy. If fosaprepitant given instead, it will be administered immediately prior to chemotherapy at 115mg IV (over 20 min). The administration site of the fosaprepitant will be noted and will be evaluated for possible venous irritation.

Dexamethasone: 20 mg orally immediately prior to chemotherapy. Ondansetron: 16 mg orally, immediately prior to the chemotherapy.

Patients agreeing to be followed on the second cycle with be assessed in the same way. During the follow-up visit after the first cycle, patients on study will be asked if they wish to continue participation during their second chemotherapy cycle (given that they are still eligible). Patients will not need to sign a separate consent, but will need to give their verbal affirmation, which will be noted in the case report form. The dosing and timing of the antiemetics may change according to the results in the first cycle, and other demographic characteristics, as follows:

Female patients:

* If there was no vomiting on the first cycle and the antiemetics were well tolerated, all antiemetics will be given identically to cycle 1.
* If any vomiting was experienced on the first cycle, patients will instead receive the typical 3-day Aprepitant (125 mg po day 1, and 80 mg po days 2 and 3), or fosaprepitant 150 mg IV (given over 30 minutes) on day 1 only. (The choice of the Aprepitant or fosaprepitant regimen will be at the discretion of the ordering oncologist). Ondansetron and dexamethasone will be given as on cycle 1. Additionally, 12mg of dexamethasone will be given on day 3

Male patients:

* For those aged 50 or older, if there was no vomiting with the first cycle and the antiemetics were well tolerated, all antiemetics will be given identically to cycle1 except that the Aprepitant dose will be reduced to one 80 mg oral administration on day 1. If fosaprepitant is used, it will be given at a total dose of 75 mg over 15 minutes. All will be given immediately prior to chemotherapy. Ondansetron and dexamethasone will be given as with cycle1.
* For those under age 50, if there was no vomiting on the first cycle and the antiemetics were well tolerated, all antiemetics will be given identically to cycle1.
* Male patients of any age, if they experienced any vomiting on the first cycle, will instead receive the typical 3-day Aprepitant (125 mg po day 1, and 80 mg po days 2 and 3), or fosaprepitant 150 mg IV (given over 30 minutes) on day 1 only. (The choice of the Aprepitant or fosaprepitant regimen will be at the discretion of the ordering oncologist). Ondansetron and dexamethasone will be given as on cycle1. Additionally, 12mg of dexamethasone will be given on day 3.

Statistics and Analysis: The investigators will compute the relevant proportions and corresponding 95% confidence interval. The association of emesis control rate by gender and other socio-demographic and clinical covariates will be examined using Chi-square test, in case of small sample size Fisher's exact test will be used. Similar analysis will be performed to examine the secondary endpoints of complete control, complete emesis control and complete nausea control in the acute emesis period (first 24 hours after chemotherapy), delayed emesis period (24 - 120 hour period after chemotherapy) and in the control in the second cycle of chemotherapy.

Justification of sample size: The investigators anticipate to recruit a total of 50 patients over one year after protocol approval, from prior experience with usage of carboplatin, the investigators expect approximately 60% will be females. The investigators project conservatively a 70% complete control rate based on prior literature (i.e. a 62% complete control rate in women and an 82% complete control rate in men). To evaluate the adequacy of the sample size (i.e. number of emesis control observed), precision was computed, as measured by the width of the 95% Confidence Interval (CI), with which the proportion of emesis control rate can be estimated. The width of the 95% CI will be no greater than 26.7% (i.e. +/-the lower and upper limit of complete control rate will be 55.4% to 82.1%) with the proposed sample size based on exact Clopper-Pearson formula.

Data and Safety Monitoring Board (DSMB) will be the primary data monitoring and safety group. Information required in reports by this committee will include 1) summaries of accrual rates and patterns; 2) information on all adverse events and protocol violations; and 3) efficacy results at the time of each DSMB meeting, which will not be available to the investigators. Note, there is no interim analysis specified for this trial. This committee will meet at least annually. The majority of the members will not be from any of the study institutions, and no member will be involved in any way with the study. Membership will include as a minimum: a statistician, a medical oncologist, and a research oncology nurse.

ELIGIBILITY:
Inclusion Criteria:

* No prior chemotherapy
* Confirmed malignancy, scheduled to receive carboplatin monotherapy, or carboplatin in combination with agents of minimal, low, or moderate emetic potential
* Laboratory parameters adequate for chemotherapy

Exclusion Criteria:

* Patients with Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 3 or 4
* Presence of nausea and vomiting or use of major antiemetic agents during the 24 hours before chemotherapy administration
* Patients receiving radiotherapy within 5 days prior to the carboplatin
* Pregnancy or lactation
* Known allergy to any of the 3 antiemetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2021-02-11 (Actual); Study Completion 2021-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Gralla, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (2):
- United States (2):
  - Jacobi Medical Center, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hesketh PJ. Chemotherapy-induced nausea and vomiting. N Engl J Med. 2008 Jun 5;358(23):2482-94. doi: 10.1056/NEJMra0706547. No abstract available. PMID 18525044
- [Background] Roila F, Herrstedt J, Aapro M, Gralla RJ, Einhorn LH, Ballatori E, Bria E, Clark-Snow RA, Espersen BT, Feyer P, Grunberg SM, Hesketh PJ, Jordan K, Kris MG, Maranzano E, Molassiotis A, Morrow G, Olver I, Rapoport BL, Rittenberg C, Saito M, Tonato M, Warr D; ESMO/MASCC Guidelines Working Group. Guideline update for MASCC and ESMO in the prevention of chemotherapy- and radiotherapy-induced nausea and vomiting: results of the Perugia consensus conference. Ann Oncol. 2010 May;21 Suppl 5:v232-43. doi: 10.1093/annonc/mdq194. No abstract available. PMID 20555089
- [Background] NCCN Guidelines, Antiemesis, Version I.2015
- [Background] Tanioka M, Kitao A, Matsumoto K, Shibata N, Yamaguchi S, Fujiwara K, Minami H, Katakami N, Morita S, Negoro S. A randomised, placebo-controlled, double-blind study of aprepitant in nondrinking women younger than 70 years receiving moderately emetogenic chemotherapy. Br J Cancer. 2013 Aug 20;109(4):859-65. doi: 10.1038/bjc.2013.400. Epub 2013 Jul 16. PMID 23860530
- [Background] Ito Y, Karayama M, Inui N, Kuroishi S, Nakano H, Nakamura Y, Yokomura K, Toyoshima M, Shirai T, Masuda M, Yamada T, Yasuda K, Hayakawa H, Suda T, Chida K. Aprepitant in patients with advanced non-small-cell lung cancer receiving carboplatin-based chemotherapy. Lung Cancer. 2014 Jun;84(3):259-64. doi: 10.1016/j.lungcan.2014.03.017. Epub 2014 Mar 27. PMID 24746177
- [Background] Yahata H, et al. Ann Oncol. 25 (Suppl 4): abstract 1481PD, 2014
- [Background] Gralla R, Jordan K, Rapoport B et al. Assessing the magnitude of antiemetic benefit with the addition of the NK1 receptor antagonist (NK1) aprepitant for all platinum agents: analysis of 1,872 patients (pts) in prospective randomized clinical phase III trials (RCTs) [abstract9057]. J Clin Oncol 2010; 28: 9057.
- [Background] Hesketh PJ, et al. Efficacy and safety of rolapitant for prevention of chemotherapy-induced nausea and vomiting (CINV) in moderately emetogenic therapy (MEC). J Clin Oncol 33 (Suppl): abstract 9622, 2015
- [Background] Navari RM, Reinhardt RR, Gralla RJ, Kris MG, Hesketh PJ, Khojasteh A, Kindler H, Grote TH, Pendergrass K, Grunberg SM, Carides AD, Gertz BJ. Reduction of cisplatin-induced emesis by a selective neurokinin-1-receptor antagonist. L-754,030 Antiemetic Trials Group. N Engl J Med. 1999 Jan 21;340(3):190-5. doi: 10.1056/NEJM199901213400304. PMID 9917226
- [Background] Roila F, Ruggeri B, Ballatori E, Fatigoni S, Caserta C, Licitra L, Mirabile A, Ionta MT, Massidda B, Cavanna L, Palladino MA, Tocci A, Fava S, Colantonio I, Angelelli L, Ciuffreda L, Fasola G, Zerilli F. Aprepitant versus metoclopramide, both combined with dexamethasone, for the prevention of cisplatin-induced delayed emesis: a randomized, double-blind study. Ann Oncol. 2015 Jun;26(6):1248-1253. doi: 10.1093/annonc/mdv132. Epub 2015 Mar 5. PMID 25743855
- [Background] Roila F, Ruggeri B, Ballatori E, Del Favero A, Tonato M. Aprepitant versus dexamethasone for preventing chemotherapy-induced delayed emesis in patients with breast cancer: a randomized double-blind study. J Clin Oncol. 2014 Jan 10;32(2):101-6. doi: 10.1200/JCO.2013.51.4547. Epub 2013 Dec 9. PMID 24323030
- [Background] Grunberg S, Chua D, Maru A, Dinis J, DeVandry S, Boice JA, Hardwick JS, Beckford E, Taylor A, Carides A, Roila F, Herrstedt J. Single-dose fosaprepitant for the prevention of chemotherapy-induced nausea and vomiting associated with cisplatin therapy: randomized, double-blind study protocol--EASE. J Clin Oncol. 2011 Apr 10;29(11):1495-501. doi: 10.1200/JCO.2010.31.7859. Epub 2011 Mar 7. PMID 21383291
- [Background] Lasseter KC, Gambale J, Jin B, Bergman A, Constanzer M, Dru J, Han TH, Majumdar A, Evans JK, Murphy MG. Tolerability of fosaprepitant and bioequivalency to aprepitant in healthy subjects. J Clin Pharmacol. 2007 Jul;47(7):834-40. doi: 10.1177/0091270007301800. Epub 2007 May 24. PMID 17525168
- [Background] Aapro M, Fabi A, Nole F, Medici M, Steger G, Bachmann C, Roncoroni S, Roila F. Double-blind, randomised, controlled study of the efficacy and tolerability of palonosetron plus dexamethasone for 1 day with or without dexamethasone on days 2 and 3 in the prevention of nausea and vomiting induced by moderately emetogenic chemotherapy. Ann Oncol. 2010 May;21(5):1083-8. doi: 10.1093/annonc/mdp584. Epub 2010 Jan 15. PMID 20080830
- [Background] Ito Y, Tsuda T, Minatogawa H, Kano S, Sakamaki K, Ando M, Tsugawa K, Kojima Y, Furuya N, Matsuzaki K, Fukuda M, Sugae S, Ohta I, Arioka H, Tokuda Y, Narui K, Tsuboya A, Suda T, Morita S, Boku N, Yamanaka T, Nakajima TE. Placebo-Controlled, Double-Blinded Phase III Study Comparing Dexamethasone on Day 1 With Dexamethasone on Days 1 to 3 With Combined Neurokinin-1 Receptor Antagonist and Palonosetron in High-Emetogenic Chemotherapy. J Clin Oncol. 2018 Apr 1;36(10):1000-1006. doi: 10.1200/JCO.2017.74.4375. Epub 2018 Feb 14. PMID 29443652
- [Background] Geling O, Eichler HG. Should 5-hydroxytryptamine-3 receptor antagonists be administered beyond 24 hours after chemotherapy to prevent delayed emesis? Systematic re-evaluation of clinical evidence and drug cost implications. J Clin Oncol. 2005 Feb 20;23(6):1289-94. doi: 10.1200/JCO.2005.04.022. PMID 15718327
- [Background] Aapro M, Rugo H, Rossi G, Rizzi G, Borroni ME, Bondarenko I, Sarosiek T, Oprean C, Cardona-Huerta S, Lorusso V, Karthaus M, Schwartzberg L, Grunberg S. A randomized phase III study evaluating the efficacy and safety of NEPA, a fixed-dose combination of netupitant and palonosetron, for prevention of chemotherapy-induced nausea and vomiting following moderately emetogenic chemotherapy. Ann Oncol. 2014 Jul;25(7):1328-1333. doi: 10.1093/annonc/mdu101. Epub 2014 Mar 5. PMID 24603643
- See also: MASCC Antiemetic tool (MAT) — http://www.mascc.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For purposes of this single arm study, the determination of whether fosaprepitant or aprepitant was administered was entirely the choice of the ordering oncologist. Both agents are NK-1 receptor antagonists. Fosaprepitant is a phosphorylated analog of aprepitant and rapidly converts to aprepitant following IV injection.
Groups:
- Low Dose Aprepitant or Fosaprepitant: In addition to standard prophylactic antiemetics (Ondansetron 16mg and Dexamethasone 20mg) patients will be given one dose of either aprepitant (125mg orally) or fosaprepitant (115mg intravenously) prior to the first cycle of carboplatin-based chemotherapy. No medications will be given afterwards
  Aprepitant 125 mg: Patient scheduled for the first cycle of carboplatin-based chemotherapy will be offered to receive low doses of either aprepitant (125mg of oral aprepitant) or 115mg of fosaprepitant intravenously for prevention of chemotherapy-induced nausea and vomiting
  Fosaprepitant 115 MG: Patient scheduled for the first cycle of carboplatin-based chemotherapy will be offered to receive low doses of either aprepitant (125mg of oral aprepitant) or 115mg of fosaprepitant intravenously for prevention of chemotherapy-induced nausea and vomiting
  Dexamethasone: Dexamethasone will be given as a part of standard CINV prophylaxis for patients receiving carboplatin-based chemotherapy, dosed at 20mg on day 1 of chemotherapy
  Ondansetron 16 MG: Ondansetron will be given as a part of standard CINV prophylaxis for patients receiving carboplatin-based chemotherapy, dosed at 16mg on day 1 of chemotherapy
Period: Overall Study
Arm/Group | Low Dose Aprepitant or Fosaprepitant
Started | 15
Completed | 13
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Ineligible | 1

BASELINE CHARACTERISTICS:
Population: For purposes of this single arm study, the determination of whether fosaprepitant or aprepitant was administered was entirely the choice of the ordering oncologist. Both agents are NK-1 receptor antagonists. Fosaprepitant is a phosphorylated analog of aprepitant and rapidly converts to aprepitant following IV injection.
Arm/Group | Low Dose Aprepitant or Fosaprepitant
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 58 [39 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Complete Control Rate of Chemotherapy-induced Nausea and Vomiting (CINV) Following 1st Cycle of Chemotherapy
Description: Complete control rate of nausea and vomiting is defined as the percentage of patients without episodes of nausea or emesis, or rescue medication administered, during the overall phase of the first carboplatin-based chemotherapy cycle. Data was collected by administration of the MASCC Antiemesis Tool. The MASCC Antiemesis Tool is an eight-item questionnaire administered to patients to assess the occurrence of vomiting and nausea both during the first 24 hours after chemotherapy as well as the occurrence of delayed nausea and vomiting from the day after to 120 hours after chemotherapy.
Time Frame: 24 hours following the first cycle of chemotherapy
Population: Data was not collected for 2 of the patients who underwent carboplatin-based chemotherapy treatment. For purposes of this single arm study, the determination of whether fosaprepitant or aprepitant was administered was entirely the choice of the ordering oncologist. Both agents are NK-1 receptor antagonists. Fosaprepitant is a phosphorylated analog of aprepitant and rapidly converts to aprepitant following IV injection.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Aprepitant or Fosaprepitant
Number analyzed (Participants) | 11
Participants
  Vomiting | 11
  Nausea | 10

2. Primary Outcome: Complete Control Rate of Chemotherapy-induced Nausea and Vomiting (CINV) Following 1st Cycle of Chemotherapy
Description: as for outcome 1
Time Frame: From 24 to 120 hours following the first cycle of chemotherapy, approximately 5 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Aprepitant or Fosaprepitant
Number analyzed (Participants) | 11
Participants
  Vomiting | 9
  Nausea | 9

3. Secondary Outcome: Complete Control Rate of Chemotherapy-induced Nausea and Vomiting (CINV) Following 2nd Cycle of Chemotherapy
Description: Complete control rate of nausea and vomiting is defined as the percentage of patients without episodes of nausea or emesis, or rescue medication administered, during overall phase of the second chemotherapy cycle. Data was collected by administration of the MASCC Antiemesis Tool. The MASCC Antiemesis Tool is an eight-item questionnaire administered to patients to assess the occurrence of vomiting and nausea both during the first 24 hours after chemotherapy as well as the occurrence of delayed nausea and vomiting from the day after to 120 hours after chemotherapy.
Time Frame: 24 hours following the second cycle of chemotherapy
Population: Only 3 participants underwent the second cycle chemotherapy treatment. For purposes of this single arm study, the determination of whether fosaprepitant or aprepitant was administered was entirely the choice of the ordering oncologist. Both agents are NK-1 receptor antagonists. Fosaprepitant is a phosphorylated analog of aprepitant and rapidly converts to aprepitant following IV injection.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Aprepitant or Fosaprepitant
Number analyzed (Participants) | 3
Participants
  Vomiting | 3
  Nausea | 3

4. Secondary Outcome: Complete Control Rate of Chemotherapy-induced Nausea and Vomiting (CINV) Following 2nd Cycle of Chemotherapy
Description: as for outcome 3
Time Frame: From 24 to 120 hours following the second cycle of chemotherapy, approximately 5 days
Population: Only 3 participants underwent the second cycle of chemotherapy treatment. For purposes of this single arm study, the determination of whether fosaprepitant or aprepitant was administered was entirely the choice of the ordering oncologist. Both agents are NK-1 receptor antagonists. Fosaprepitant is a phosphorylated analog of aprepitant and rapidly converts to aprepitant following IV injection.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Aprepitant or Fosaprepitant
Number analyzed (Participants) | 3
Participants
  Vomiting | 3
  Nausea | 3

ADVERSE EVENTS:
Time Frame: Up to 120 hours following the first and second cycle of chemotherapy. Each cycle of chemotherapy is approximately 5 days in duration. Participants were monitored for adverse events up to a total of 2 weeks in aggregate.
Description: For purposes of this single arm study, the determination of whether fosaprepitant or aprepitant was administered was entirely the choice of the ordering oncologist. Both agents are NK-1 receptor antagonists. Fosaprepitant is a phosphorylated analog of aprepitant and rapidly converts to aprepitant following IV injection.
Arm/Group | Low Dose Aprepitant or Fosaprepitant
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 1/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Aprepitant or Fosaprepitant (N=13)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Hiccoughs

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-28): https://cdn.clinicaltrials.gov/large-docs/11/NCT03237611/Prot_SAP_000.pdf